CLINICAL TRIAL: NCT01271049
Title: A Double-blind, Randomized, Controlled Evaluation of the Tolerability of a Proprietary Oil Blend in Adults Residing in Areas Endemic for Helminth Infections.
Brief Title: An Evaluation of a Novel Food Product in Adults Residing in an Area Endemic for Helminths
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to a business decision to stop the project, the study was terminated early.
Sponsor: Mondelēz International, Inc. (Industry)
Collaborators: TyraTech Technology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ABS-00-02
Record Dates: First submitted 2011-01-03; First posted 2011-01-06 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Helminthiasis
MeSH Terms: conditions — Helminthiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Food Product (Placebo Comparator): Consumption of placebo food product
  Interventions: Other: Control Food Product
- Novel Food Product (Experimental): Consumption of novel food product
  Interventions: Other: Novel Food Product

INTERVENTIONS:
Other: Novel Food Product — Novel food product containing essential oil blend
  Arms: Novel Food Product
Other: Control Food Product — Control food product
  Arms: Control Food Product

SUMMARY:
The prevalence of intestinal helminths is worldwide. This study will evaluate the tolerability of a novel food product consumed by adults residing in an area endemic for helminths.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or Female adults, age 18-45 years old inclusive on date of screening
* Showing presence of no or mild-moderate helminths

Exclusion Criteria:

* Presence of heavy helminth load
* Pregnant or lactating
* Hepatosplenomegaly or clinically significant abnormal hemoglobin, LAT or creatinine

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Measure of Safety and Tolerability using the Reactogenicity Questionairre | 43 days
  Reactogenicity will be assessed using a structured questionnaire on days 2, 14, 28, and 42 of the study. In addition, blood will be collected on study days 14 and 42 for assessment of basic hematologic and clinical chemistry parameters.

CONTACTS AND LOCATIONS:
Overall Officials: David Diemert, MD, FRCP(C), Principal Investigator — Rene Rachou Research Center, Brazil
Locations (1):
- Centro de Pesquisas Rene Rachou-FIOCRUZ, Minas Gerais, Brazil